CLINICAL TRIAL: NCT00560521
Title: Effect of Continuous Positive Airway Pressure on Fluid Absorption Among Patients With Pleural Effusion Due to Tuberculosis
Brief Title: Continuous Positive Airway Pressure on Tuberculosis Pleural Effusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Oliveira-1
Record Dates: First submitted 2007-11-16; First posted 2007-11-19 (Estimated); Last update posted 2007-11-19 (Estimated); Status verified 2007-11

CONDITIONS: Tuberculosis; Pleural Effusion
Keywords: CPAP; Tuberculosis; Pleural effusion; Physiotherapy
MeSH Terms: conditions — Tuberculosis; Pleural Effusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Active Comparator)
  Interventions: Behavioral: CPAP

INTERVENTIONS:
Behavioral: CPAP — Frequency of three times a week, using a positive end expiratory pressure (PEEP) of 10 mmH2O for 30 minutes for four weeks.

SUMMARY:
Tuberculosis (TB) remains as an important public health problem worldwide. Pleural tuberculosis is the most prevalent form of extrapulmonary presentation in immunocompetent patients.

The volume of effusion in the pleural space of patients with pleural TB may cause complications like restrictive ventilator lung functional disturb and/or pleural thickening. The respiratory physiotherapy can be adjuvant on treatment of pleural effusion tuberculosis throughout of various treatment technique.

The Continuous positive airway pressure (CPAP) is utilized in various pathologic, this improves lung mechanics by recruiting atelectatic alveoli, improving pulmonary compliance, and reducing the work of breathing.

The aim of this study is to determine the effect of CPAP on fluid absorption among patients with pleural effusion due tuberculosis.

DETAILED DESCRIPTION:
This randomized and controlled trial compared the reduction of the pleural effusion volume of the group of patients using the anti-TB standard regimen to that using the anti-TB standard regimen AND adjuvant treatment of physical therapy during four weeks.

* Control group: The patients received rifampicin, isoniazid and pyrazinamide daily(anti-TB standard regimen)
* Interventional group: The patients received anti-tb standard regime and Continuous Positive Airway Pressure (CPAP) 3 times a week for 30 minutes with positive expiratory end pressure of 10 cmH2O.

Evaluation of the pleural effusion size: a helicoidal thoracic computed tomography (CT) was carried out in all patients enrolled. The valuation was conducted by two radiologists blinded for the treatment used, specifically trained for the purpose of the study.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of pleural tuberculosis.
* Patients 18 years of age and older.

Exclusion criteria:

* Be under previous treatment of respiratory physiotherapy.
* Irregular use or abandonment of the anti-TB standard regimen.
* To fail one or more physiotherapy section.
* To fail one or more radiological evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-03; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Evaluate of pleural effusion volume | one month

CONTACTS AND LOCATIONS:
Overall Officials: Juliana F Oliveira, MD, Principal Investigator — Universidade Federal do Rio de Janeiro; Marcus B. Conde, PhD, Principal Investigator — Universidade Federal do Rio de Janeiro; Rosana S. Rodrigues, MD, Study Chair — Universidade Federal do Rio de Janeiro; Sara L. Menezes, PhD, Principal Investigator — Universidade Federal do Rio de Janeiro; Ana L. Boechat, MD, Study Chair — Universidade Federal do Rio de Janeiro; Fernanda C. Mello, PhD, Principal Investigator — Universidade Federal do Rio de Janeiro
Locations (1):
- Clementino Fraga Filho University Hospital- Federal University of Rio de Janeiro, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Background] Valdes L, Alvarez D, San Jose E, Penela P, Valle JM, Garcia-Pazos JM, Suarez J, Pose A. Tuberculous pleurisy: a study of 254 patients. Arch Intern Med. 1998 Oct 12;158(18):2017-21. doi: 10.1001/archinte.158.18.2017. PMID 9778201
- [Background] Masip J. Non-invasive ventilation. Heart Fail Rev. 2007 Jun;12(2):119-24. doi: 10.1007/s10741-007-9012-7. PMID 17492379
- [Background] Seiscento M, Conde MB, Dalcolmo MM. [Tuberculous pleural effusions]. J Bras Pneumol. 2006;32 Suppl 4:S174-81. doi: 10.1590/s1806-37132006000900003. Portuguese. PMID 17273621
- [Background] Conde MB, Loivos AC, Rezende VM, Soares SL, Mello FC, Reingold AL, Daley CL, Kritski AL. Yield of sputum induction in the diagnosis of pleural tuberculosis. Am J Respir Crit Care Med. 2003 Mar 1;167(5):723-5. doi: 10.1164/rccm.2111019. PMID 12598215
- [Result] Vandevenne A, Moyses B, Weitzenblum E, Carloz I, Methlin G. [Regional pulmonary function in unilateral sero-fibrinous pleural effusions and changes under the influence of treatment (author's transl)]. Poumon Coeur. 1981;37(3):223-8. French. PMID 7301718
- [Result] Ferrer J. Pleural tuberculosis. Eur Respir J. 1997 Apr;10(4):942-7. PMID 9150338
- [Result] Zhou A, Guo L, Tang L. Effect of an intrathoracic injection of sodium hyaluronic acid on the prevention of pleural thickening in excess fluid of tuberculous thoracic cavity. Clin Exp Pharmacol Physiol. 2003 Mar;30(3):203-5. doi: 10.1046/j.1440-1681.2003.03804.x. PMID 12603352
- [Derived] Oliveira JF, Mello FC, Rodrigues RS, Boechat AL, Conde MB, Menezes SL. Effect of continuous positive airway pressure on fluid absorption among patients with pleural effusion due to tuberculosis. Rev Bras Fisioter. 2010 Mar-Apr;14(2):127-32. doi: 10.1590/s1413-35552010005000001. Epub 2010 Apr 30. PMID 20464170